CLINICAL TRIAL: NCT00242840
Title: A 24 Week Phase IIIb/IV Single Arm Open Label Observational Study to Explore the Efficacy of Protease Inhibitors Given in Combination With Reverse Transcriptase Inhibitors to HIV-1 Infected Subjects With Protease Mutations Selected During Therapy With GW433908 Containing Antiretroviral Therapy
Brief Title: Observational Study Of A Protease Inhibitor (PI) Containing Regimen In Subjects With PI Mutations Selected During Prior Treatment With GW433908 (Fosamprenavir)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: APV30007
Record Dates: First submitted 2005-10-19; First posted 2005-10-21 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Infection, Human Immunodeficiency Virus I; HIV Infection
Keywords: protease inhibitor; ritonavir; GW433908; HIV-1; fosamprenavir
MeSH Terms: conditions — Infections; HIV Infections | interventions — Observation

INTERVENTIONS:
Drug: No intervention; Observational study

SUMMARY:
This study will assess the efficacy of subsequent protease inhibitor (PI)-containing therapy in subjects who have acquired HIV-1 protease mutations whilst receiving a GW433908 (fosamprenavir)-containing regimen.

ELIGIBILITY:
Inclusion criteria:

* Prior participation in study APV30005 AND one of the following studies: APV30001, APV30002, AZL30006, APV30003.
* Must be failing virologically (>1000 copies at two consecutive time-points) and have a screening genotype with evidence of at least one new APV-associated protease mutation: V32I (+/- I47V), I50V, I54L/M, I84V acquired since commencing treatment with GW433908.

Exclusion criteria:

* Have 2 or more of the primary resistance mutations D30N, G48V, V82A/F/T/S and L90M.
* Have a medical need for use of an non-nucleoside reductase transferase inhibitor (NNRTI).
* Have an acute CDC Class C event requiring therapeutic intervention.
* Are pregnant or lactating.
* Have any other condition which in the opinion of the investigator would preclude their participation.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-06; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (6):
- United States (5):
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Augusta, Georgia
- GSK Investigational Site, Brescia, Lombardy, Italy